CLINICAL TRIAL: NCT00218283
Title: Treatment of Smokeless Tobacco Users
Brief Title: Nicotine Lozenge to Reduce Smokeless Tobacco Use
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: University of Minnesota (Other)
Responsible Party: Dorothy Hatsukami, University of Minnesota
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIDA-14404-3; R01-14404-3; DPMC
Record Dates: First submitted 2005-09-16; First posted 2005-09-22 (Estimated); Last update posted 2017-01-10 (Estimated); Status verified 2008-06

CONDITIONS: Tobacco Use Disorder
Keywords: Nicotine Dependence; Tobacco Dependence
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Tobacco Use Cessation Devices; Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 - Nicotine Lozenge (Experimental): Use of nicotine lozenge plus behavioral counseling to help reduce tobacco use prior to quit date.
  Interventions: Drug: Nicotine Lozenge
- 2 Behavioral counseling (Placebo Comparator): Use of behavioral counseling alone to help reduce tobacco use prior to quit date.
  Interventions: Behavioral: Behavioral Counseling

INTERVENTIONS:
Drug: Nicotine Lozenge — Oral Nicotine replacement product
  Other Names: Commite Nicotine lozenge
  Arms: 1 - Nicotine Lozenge
Behavioral: Behavioral Counseling — Use of behavioral counseling to reduce tobacco use.
  Arms: 2 Behavioral counseling

SUMMARY:
Smokeless tobacco (ST), which includes both chewing tobacco and snuff, has as many health risks associated with its use as cigarettes. While there are many treatment programs that focus on stopping tobacco use, there are no interventions that specifically focus on reducing tobacco use. This study will evaluate the effectiveness of nicotine lozenge at reducing tobacco use in ST users.

DETAILED DESCRIPTION:
Individuals who use ST are at risk for developing heart disease, stroke, high blood pressure, and cancer. Other long-term effects include tooth abrasion, gum recession, and loss of bone in the jaw. Many individuals who use ST recognize the health risks associated with ST, but either do not want to quit or feel that it is impossible to quit. For these individuals, tobacco reduction may be an important transitional goal, either prior to quitting or as a treatment endpoint. The need exists for a program specifically aimed towards reducing, rather than quitting, tobacco use. The purpose of this study is to evaluate the effectiveness of nicotine gum at reducing ST use, as well as assessing the motivation to either quit or sustain lower levels of ST use.

This 8-week study will enroll frequent users of ST. Participants will be randomly assigned to receive either nicotine lozenge plus behavioral counseling or behavioral counseling alone. All participants will be asked to alternate use of their usual ST brand with nicotine lozenge or placebo in order to reduce nicotine intake by 50% during the first 4 weeks and by 75% the following 4 weeks. Participants will be required to maintain a daily tobacco use diary. Study visits will occur once a week. Tobacco levels will be monitored with urine tests, and questionnaires will be completed to assess tobacco use. Follow-up evaluations will occur 12 and 26 weeks following the end of treatment.

ELIGIBILITY:
Inclusion Criteria:

* No interest in stopping ST use within 90 days of study entry
* Using ST at least 6 times a day in the 6 months prior to study entry
* Willing to use contraception throughout the study

Exclusion Criteria:

* Current use of tobacco or nicotine products, other than ST
* Current unstable medical condition
* Use of any medication that may affect tobacco use or be affected by a reduction in tobacco use
* Meets DSM-IV diagnostic criteria for any psychiatric disorder or substance abuse disorder within 6 months of study entry
* Use of any psychotropic medication within 6 months of study entry
* Pregnant or breastfeeding

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2005-01; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Reduction in tobacco use (measured by tobacco daily diary at Week 8, and the 12- and 26-week follow-up evaluations) | 8, 12 and 26 weeks
Toxicity profile of carcinogen metabolites (measured by urine screens at Week 8, and the 12- and 26-week follow-up evaluations) | 8, 12 and 26 weeks
Number of unsuccessful attempts to quit using tobacco (measured by tobacco use questionnaire at Week 8, and the 12- and 26-week follow-up evaluations) | 8, 12 and 26 weeks
Abstinence from tobacco (measured by tobacco use questionnaire at Week 8, and the 12- and 26-week follow-up evaluations) | 8, 12 and 26 weeks

SECONDARY OUTCOMES:
Motivation and self-efficacy (measured by a questionnaire at Week 8, and the 12- and 26-week follow-up evaluations) | 8, 12 and 26 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dorothy Hatsukami, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States